CLINICAL TRIAL: NCT06668207
Title: Evaluation of the Effect of Carbohydrate Quality on Physical Activity Enjoyment and Burnout in Athletes
Brief Title: Carbohydrate Quality and Its Impact on Athletic Enjoyment and Burnout
Status: Completed | Type: Observational
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Emine Elibol, Assist. Prof., Ankara Yildirim Beyazıt University
Other Study IDs: AYBUELİBOL003
Record Dates: First submitted 2024-10-23; First posted 2024-10-31 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-06

CONDITIONS: Athlete
Keywords: Carbohydrate quality; sport; physical activity; burnout
MeSH Terms: conditions — Motor Activity; Burnout, Psychological

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- adult athletes: This study aimed to evaluate the effect of carbohydrate quality on enjoyment of physical activity and burnout in athletes. Data were collected from 139 active athletes aged 19 to 35 years using a Demographic Structure Questionnaire, the Athlete Burnout Questionnaire (ABQ), and the Physical Activity Enjoyment Scale (PACES). Carbohydrate quality was assessed using food frequency data, and the results were analyzed with SPSS 24 software.

SUMMARY:
This study aimed to evaluate the effect of carbohydrate quality on enjoyment of physical activity and burnout in athletes. Data were collected from 139 active athletes aged 19 to 35 years using a Demographic Structure Questionnaire, the Athlete Burnout Questionnaire (ABQ), and the Physical Activity Enjoyment Scale (PACES). Carbohydrate quality was assessed using food frequency data, and the results were analyzed with SPSS 24 software.

DETAILED DESCRIPTION:
Objective: The aim of this study was to evaluate the effect of carbohydrate quality on enjoyment of physical activity and burnout in athletes.

Method: A total of 139 active athletes aged 19 to 35 years participated in the study. Participants completed a Demographic Structure Questionnaire, the Athlete Burnout Questionnaire (ABQ), and the Physical Activity Enjoyment Scale (PACES). To assess carbohydrate quality, food frequency data were collected, and scores were based on fiber intake, the whole-to-total grain ratio, glycemic index, and solid-to-total carbohydrate ratio, each evaluated on a scale from 1 to 5 points. The resulting scores were categorized into five quartiles, with Q5 indicating the highest and Q1 the lowest carbohydrate quality. Data were analyzed using SPSS 24 software.

ELIGIBILITY:
Inclusion Criteria:

* Only athletes who are actively participating in sports
* Age range of 19 to 35 years
* Voluntary participation

Exclusion Criteria:

-Individuals engaging in irregular physical activity

Ages: 19 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community sample in Ankara, Turkey
Sampling Method: Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Evaluating carbohydrate quality | Basaline
  A total of 132 food groups obtained from the food consumption frequency questionnaire were analyzed. Daily intake (g/day) was calculated using the BeBiS program with a global database, considering the amount and frequency of food consumed by each participant. Glycaemic Index (GI) values were also determined using the BeBiS program, taking into account the amount and frequency of food consumed. To determine the Carbohydrate Quality Index score, each of the four components (fiber intake, whole grain ratio, glycaemic index, and total carbohydrate ratio) was evaluated on a scale from 1 to 5 points. The scores for each component were then summed. Q5 indicates the highest and Q1 indicates the lowest carbohydrate quality.

SECONDARY OUTCOMES:
Athlete Burnout Questionnaire (ABQ) | Basaline
  The Athlete Burnout Questionnaire was used to determine the level of burnout in athletes. The scale consists of 13 questions scored on a five-point Likert scale (1-Never, 2-Sometimes, 3-Often, 4-Frequently, 5-Always) and is divided into three subdimensions: "Decreased Sense of Achievement," "Emotional/Physical Exhaustion," and "Depersonalization." The total score can range from 15 to 65, with higher scores indicating higher levels of burnout.
Physical Activity Enjoyment Scale (PACES) | Basaline
  The Physical Activity Enjoyment Scale (PACES) was used to assess the level of enjoyment athletes experience during physical activity. The scale consists of 8 questions scored on a scale from 1 to 7, with a maximum score of 56 and a minimum score of 8. Higher scores indicate greater enjoyment of physical activity.
Sociodemographic characteristics | Basaline
  Sociodemographic characteristics will be assessed using a structured questionnaire developed by the researchers. The questionnaire will include items measuring age, gender, education level, and income status. The results will be presented as numbers and percentages for each characteristic
Body Mass Index (BMI) | Basaline
  Kilograms per square meter (kg/m2)
Body weight | Basaline
  Body weight in kg
Height | Basaline
  Height in cm

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yıldırım Beyazıt University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No